CLINICAL TRIAL: NCT06278428
Title: Genotype, Phenotype, and Disease Progression of Developmental Epileptic Encephalopathy With Onset Before 2 Years of Age
Status: Recruiting | Type: Observational
Sponsor: Number 2 Children's Hospital, Ho Chi Minh City (Other)
Responsible Party: Principal Investigator, Thuy-Minh-Thu NGUYEN, Principal Investigator, Number 2 Children's Hospital, Ho Chi Minh City
Other Study IDs: DEE UMC
Record Dates: First submitted 2024-02-19; First posted 2024-02-26 (Actual); Last update posted 2025-01-09 (Actual); Status verified 2025-01

CONDITIONS: Epilepsy; Seizure; Child Development; Gene Abnormality; Early Onset Disorder
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Biospecimen Retention: Samples With DNA — blood
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- early onset developmental epileptic encephalopathy: Select one that meets all 5 of the following criteria:
  1. Diagnosed with EIDEE or EIMFS or ISS or SMEI or EMAS (according to ILAE's diagnostic criteria 2022)
  2. Diagnosed with drug-resistant epilepsy according to ILAE 2010 criteria (according to ILAE's diagnostic criteria 2010)
  3. Age at the start of participating in the study ranged from 0 to 23 months old
  4. Relatives agree to participate in the research
  5. There is no medical history of any diagnosis of hypoxic encephalopathy or inflammatory encephalopathy or traumatic encephalopathy or cerebral infarction or cerebral hemorrhage.

SUMMARY:
According to estimates by the World Health Organization in 2019, more than 50 million people around the world have epilepsy. Nearly 80% of patients with epilepsy live in developing countries. Among them, children under 2 years old are the group with the highest incidence of epilepsy, and at the same time, the most dangerous epilepsy groups are also likely to start at these ages. World medical literature on epileptic encephalopathy and early-onset development before 2 years of age records that 71% of children have severe intellectual disability and 60% of children show signs of autism spectrum disorder, of which Children with epileptic and developmental encephalopathy due to genetic causes are at higher risk of developing neurodevelopmental disorders than children with epileptic and developmental encephalopathy due to other causes. However, in Vietnam, there is no research on this topic.

The question is what are the phenotypes, genotypes, and progression after 2 years of follow-up of Vietnamese children with epileptic and developmental encephalopathy with onset before 2 years of age?

DETAILED DESCRIPTION:
According to estimates by the World Health Organization in 2019, more than 50 million people around the world have epilepsy. Nearly 80% of patients with epilepsy live in developing countries. In Vietnam, the incidence of epilepsy is approximately 40 per 100,000 per year. The incidence of the disease in children is higher than in adults. Among them, children under 2 years old are the group with the highest incidence of epilepsy, and at the same time, the most dangerous groups of epilepsy are also likely to start at these ages, such as West syndrome, Dravet syndrome, and Dravet syndrome. Ohtahara syndrome. These syndromes belong to the group of epileptic and developmental encephalopathies. This group of diseases can be caused by many causes, such as structural, metabolic, infectious, and genetic causes. However, in children and young people, genetic causes are more common.

Thanks to the development of biotechnology and genetics, medicine is now discovering more and more genes related to epilepsy syndromes that begin before 2 years of age, which helps choose treatment methods for the disease. causes of epilepsy such as using the keto diet in children with loss-of-function mutations in SLC2A1 or avoiding sodium channel blockers in children with Dravet syndrome due to loss-of-function mutations in SCN1A. In addition, children with epileptic and developmental encephalopathy due to genetic causes are also at higher risk of global developmental delay and autism spectrum disorders. Therefore, monitoring the progress of children with epileptic and developmental encephalopathy due to genetic causes plays an important role in early intervention, helping to improve disease prognosis.

World medical literature on epileptic encephalopathy and early-onset development before 2 years of age records that 71% of children have severe intellectual disability and 60% of children show signs of autism spectrum disorder, of which Children with epileptic and developmental encephalopathy due to genetic causes are at higher risk of developing neurodevelopmental disorders than children with epileptic and developmental encephalopathy due to other causes. In our country, there have been a number of studies on epileptic and developmental encephalopathy, as follows: A study conducted at Children's Hospital 2 showed the detection rate of gene mutations in patients with epileptic encephalopathy. menstruation and development is 38%, mainly SCN1A genotype mutation and Dravet syndrome phenotype. Another study that followed the short-term course of epileptic and developmental encephalopathy patients on the keto diet found that the majority of Dravet syndrome patients responded well to this treatment. However, studies in our country only describe genotypes and phenotypes separately without including progression, or only monitor the progression of phenotypes with treatment methods without paying attention to genotypes, or do not focus on focuses on studying the group of epileptic and developmental encephalopathies with onset before 2 years of age, which is the group with the highest incidence and most danger. Furthermore, most studies are cross-sectional or only monitor short-term progress. Therefore, the question is what is the phenotype, genotype, and progression after 2 years of follow-up of children with epileptic and developmental encephalopathy with onset before 2 years of age? We want to conduct this study to answer the above question.

Researching this issue will make an important contribution to a better understanding of the genotype, phenotype, and course of epileptic and developmental encephalopathies, thereby aiding the treatment and management of the disease.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed with Early infantile developmental and epileptic encephalopathy or Epilepsy of infancy with migrating focal seizures or infantile spasms syndrome or severe myoclonic epilepsy of infancy or Epilepsy with myoclonic-atonic seizures
2. Diagnosed with drug-resistant epilepsy according to ILAE 2010 criteria
3. Age at the start of participating in the study ranged from 0 to 23 months old
4. Relatives agree to participate in the research
5. There is no medical history of any diagnosis of hypoxic encephalopathy or inflammatory encephalopathy or traumatic encephalopathy or cerebral infarction or cerebral hemorrhage.

Exclusion Criteria:

Patients were removed from the study when they were lost to follow-up at 6 months

-

Max Age: 23 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The study population was patients with severe, early-onset epilepsy, suspected of having a genetic etiology
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-02-27 (Actual); Primary Completion 2028-11-01 (Estimated); Study Completion 2028-11-01 (Estimated)

PRIMARY OUTCOMES:
Genotye of early-onset developmental epileptic encephalopathy | 2/2024- 4/2025
  Describing the genotype of early-onset developmental epileptic encephalopathy

OTHER OUTCOMES:
Phenotye of early-onset developmental epileptic encephalopathy | 2/2024-4/2025
  Describing the phenotype of early-onset developmental epileptic encephalopathy
Progression of epileptic encephalopathy and early onset developmental epileptic encephalopathy | 4/2025-4/2027
  Describing the progression of epileptic encephalopathy and early onset developmental epileptic encephalopathy

CONTACTS AND LOCATIONS:
Locations (2):
- Vietnam (2):
  - Children hospital number 2, Ho Chi Minh City
  - University of Medicine and Pharmacy at Ho Chi Minh city, Ho Chi Minh City

IPD SHARING:
Plan to Share IPD: Undecided